CLINICAL TRIAL: NCT00938119
Title: The Care China-Diabetes Registry A 12-month, Multi-centre, Prospective, Observational Registry Study to Investigate the Efficacy and Safety of CYPHER Select TM+ Sirolimus-eluting Coronary Stent Among Chinese Diabetic Patients With Coronary Artery Disease in Routine Clinical Practice
Brief Title: Care China-Diabetes
Status: Terminated | Type: Observational
Why Stopped: the product was delisted.
Sponsor: Johnson & Johnson Medical, China (Industry)
Responsible Party: Sponsor
Other Study IDs: CDS-200801
Record Dates: First submitted 2009-06-24; First posted 2009-07-13 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2011-07

CONDITIONS: Cardiovascular Disease; Diabetes
Keywords: Cardiovascular disease; Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Diabetes patient
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetes patients with PCI: this is single group

SUMMARY:
This multicenter, prospective, observational registry will assess efficacy and safety outcomes associated with percutaneous coronary intervention (PCI) with implantation of the CYPHER Select™+ Sirolimus-eluting Coronary Stents in Chinese diabetic patients with coronary artery disease in routine clinical practice.

DETAILED DESCRIPTION:
The study objective is to assess the incidences of major adverse cardiovascular events (MACE; defined as a composite of clinically driven target-lesion revascularization, cardiac death, any myocardial infarction, and stent thrombosis) at 12-month follow-up, and of stent thrombosis at 1-day, and 1- and 12-month follow-up. Pre-specified analyses will be performed among patient subpopulations according to level of glycemic control (HbA1c level < 6.5% or > 6.5%); reference vessel diameter by quantitative coronary angiography (< 2.5 mm and > 2.5 mm); and stented length (8-18 mm; 23-33 mm; and >33 mm). Quantitative coronary angiographic (QCA) analysis will be performed at the core lab of the China Cardiovascular Research Foundation for all pre- and post-index procedure angiograms and during the 12-month follow-up period for the pre- and post-reintervention procedures in those cases of clinically-driven PCI revascularization. Also, multivariable analyses will be conducted to investigate potential predictors of 12-month MACE rate in routine clinical practice.

The registry will be conducted at about 45 centers in China, where the CYPHER Select™+ Sirolimus-eluting Coronary Stent is commercially available. Data will be collected on 2,500 diabetic patients treated with the CYPHER Select™ + Sirolimus-eluting Coronary Stent only.

Primary outcome: MACE (clinically driven TLR, cardiac death, MI, ST) at 12 months Secondary outcome: ARC (probable + definite) ST at 1-day, and 1 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 80 (inclusive) receiving CYPHER SELECT™+ Sirolimus-eluting Coronary Stent according to standard clinical practice when financially feasible
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.
* Patient has diagnosis of diabetes or is diagnosed with it before or during the index procedure hospitalization based on disease diagnosis criteria

Exclusion Criteria:

* Any contraindication to any of the following medications: aspirin, heparin, thienopyridines (clopidogrel/ticlopidine), stainless steel, contrast agents, or sirolimus
* An elective surgical procedure is planned that would necessitate interruption of antiplatelet drugs during the first 6 months post enrollment
* Cardiogenic shock
* Terminal illness with life expectancy <1 year
* ST-segment elevation myocardial infarction within 7 days prior to the index procedure
* Any patient who received coronary stent(s) within 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will be conducted at approximately 45 centers in China where the CYPHER SelectTM+ Sirolimus-eluting Coronary Stent is commercially available. Data will be collected on 2,500 diabetic patients treated only with the CYPHER Select™+ Sirolimus-eluting Coronary Stent during the index procedure. Enrolled diabetic patients are confirmed and diagnosed with Diabetes before or during the index procedure hospitalization, i.e., those receiving active treatment with an oral hypoglycemic agent or insulin, patients with diagnosis of diabetes who were on dietary therapy alone or patients with an abnormal blood glucose level after an overnight fast as defined by local standards.
Sampling Method: Probability Sample
Enrollment: 1603 (Actual)
Dates: Start 2009-08; Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
MACE (clinically driven TLR, cardiac death, MI, ST) at 12 months | 12 months

SECONDARY OUTCOMES:
ARC (probable + definite) ST at 1-day, and 1 and 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yue Jin, MD, Phd, Principal Investigator — Cardiovascular Institute & Fu Wai Hospital; Lv Shu Zheng, MD, Principal Investigator — Beijing Anzhen Hospital of the Capital University of Medical Sciences; Chen Yun Dai, MD, Phd, Principal Investigator — Chinese PLA General Hospital; Wang Le feng, Principal Investigator — Beijing Chaoyang Hospital Affiliated to the Capital University of Medical Sciences; Gao Wei, MD, Phd, Principal Investigator — Peking University Third Hospital; Wang Wei Min, MD, PhD, Principal Investigator — Peking University People's Hospital; Huo Yong, MD, PhD, Principal Investigator — Peking University First Hospital; Fang Quan, MD, PhD, Principal Investigator — Peking Union Medical College Hospital; He Qing, MD, PhD, Principal Investigator — Beijing Hospital; Liu Hui Liang, MD, Principal Investigator — General Hospital of Armed Police Forces; Li Hui, MD, Principal Investigator — General Hospital of Daqing Oilfield; Chen Ji Yan, MD, PhD, Principal Investigator — Guangdong Provincial People's Hospital; Du Zhi Min, MD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Hou Yu Qing, MD, Principal Investigator — Southern Medical University, China; Li Wei Min, MD, Principal Investigator — First Affiliated Hospital of Harbin Medical University; Yu Bo, MD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University; Fu Guo Sheng, MD, Principal Investigator — Sir Run Run Shaw Hospital Affiliated with School of Medicine,Zhejiang University; Wang Jian An, MD, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Zhu Jian Hua, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University College of Medicine; Liu Bin, MD, Principal Investigator — The Second Affiliated Hospital of Jilin University; Cui Lian Qun, MD, PhD, Principal Investigator — Shandong Provincial Hospital; Zhang Zheng, MD, PhD, Principal Investigator — Lanzhou University First Hospital; Chen Shao Liang, MD, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Xu Biao, MD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Li Lang, MD, PhD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University; Ge Jun Bo, MD, PhD, Principal Investigator — Fudan University; He Ben, MD,PhD, Principal Investigator — Shanghai Jiaotong University School of Medicine affiliated Renji Hospital; Shen Wei Feng, MD, PhD, Principal Investigator — Shanghai Jiaotong University School of Medicine affiliated Ruijin Hospital; Xu Ya Wei, MD, PhD, Principal Investigator — Shanghai Tenth People's Hospital of Tongji University; Han Ya Ling, MD, PhD, Principal Investigator — General Hospital of Shenyang Military Region; Pang Wen Yue, MD, PhD, Principal Investigator — Shengjing Hospital; Li Bao, MD,PhD, Principal Investigator — Shanxi Cardiovascular Hospital; Lv Ji Yuan, MD, Principal Investigator — The First Affiliated Hospital of Shanxi Medical University; Liu Yin, MD, PhD, Principal Investigator — Tian Jin Chest Hospital; Qi Xiang Qian, MD, Principal Investigator — TEDA International Cardiovascular Hospital; Jiang Tie Min, MD, Principal Investigator — The Affiliated Hospital of Medical College of Chinese Armed Police Forces; Lu Cheng Zhi, MD, Principal Investigator — Tianjin First Central Hospital; Huang Wei Jian, MD, PhD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University; Sun Ying Xian, MD, Principal Investigator — First Hospital of China Medical University; Li Guo Qing, MD, Principal Investigator — People's Hospital of Xinjiang Uygur Autonomous Region; Yuan Zu Yi, MD, Principal Investigator — The First Hospital of Xian Jiao Tong University; Wang Hai Chang, MD, Principal Investigator — Xijing Hospital; Wang Yan, MD,PhD, Principal Investigator — Zhongshan Hospital Xiamen University; Gao Chuan Yu, MD, PhD, Principal Investigator — Henan Provincial People's Hospital; Wang Chun, MD, PhD, Principal Investigator — Peking University, Shen Zhen Hospital; Yong Wang, MD, PhD, Principal Investigator — China-Japan Friendship Hospital
Locations (46):
- China (46):
  - Beijing Anzhen Hospital of the Capital University of Medical Science, Beijing, Beijing Municipality
  - General Hospital of Armed Police Forces, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality
  - Xuan Wu Hospital Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijng, Beijing Municipality
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Lanzhou University First Hospita, Lanzhou, Gansu
  - Peking University, Shenzhen Hospital, Guangdong, Guangdong
  - NanFang Hospital Affiliated to Southern Medical University, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital,Sun Yat-Sen University, Guangzhou, Guangdong
  - Peace Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Jilin University, Changchun, Jilin
  - The General Hospital of Shenyang Military Command, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Hospital Of Medical College Qingdao University, Qingdao, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Jiaotong University School of Medicine affiliated Renji Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xijing Hospital, Xian, Shanxi
  - Tian Jin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Center Hospital, Tianjin, Tianjin Municipality
  - People's Hospital Of XinJiang Uygur Autonomous Region, Urumuqi, Xinjiang
  - Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - Cardiovascular Institute & Fu Wai Hospital, Beijing
  - General Hospital of Daqing Oilfield, Daqing
  - Sir Run Run Shaw Hospital, Hangzhou
  - Shandong Provincial Hospital, Jinan
  - Shanghai Tenth People's Hospital of Tongji University, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Teda International Cardiovascular Hospital, Tianjin
  - The Affiliated Hospital of Medical College of Chinese Armed Police Forces, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou
  - The First Hospital of Xian Jiao Tong University, Xi'an